CLINICAL TRIAL: NCT01151423
Title: A Phase II, Single-blind, Randomized, Placebo-controlled Trial to Study the Efficacy and Safety of Anti-von Willebrand Factor Nanobody Administered as Adjunctive Treatment to Patients With Acquired Thrombotic Thrombocytopenic Purpura
Brief Title: Study to Assess Efficacy and Safety of Anti-von Willebrand Factor (vWF) Nanobody in Patients With Acquired Thrombotic Thrombocytopenic Purpura (aTTP)
Acronym: TITAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALX0681-2.1/10; 2010-019375-30 (EudraCT Number)
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2019-05

CONDITIONS: Acquired Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — caplacizumab

STUDY DESIGN:
Who Masked: Participant
Masking Description: A single-blinded study design was initiated because, in the initial versions of the protocol, the dosing regimen could be adjusted dependent on the results of the Ristocetin Cofactor (RICO) test following the initial dose. Therefore, a double-blind design was not feasible because the results of the RICO test effectively unblinded the Investigator. Single-blind design was maintained due to the objective nature of the primary endpoint.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caplacizumab (Experimental): Caplacizumab 10 mg once daily
  Interventions: Biological: Caplacizumab
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Caplacizumab — * Subjects received a first intravenous (i.v.) bolus of 10 mg (filled at 5 mg/mL) caplacizumab via push injection within 6 hours to 15 minutes prior to the first PE on study. The first PE on study could either be the very first PE session for the current episode of aTTP (if the subject was randomized prior to the initiation of PE) or the second PE session (if the subject was randomized after a single PE session).
  * The first PE on study was followed by subcutaneous (s.c.) administration of 10 mg study drug within 30 minutes after the end of the PE procedure.
  * All subsequent study drug administrations were daily s.c. injections within 30 minutes after the end of the PE procedure (if applicable) or within 24 hours of the previous dose.
  * Subjects received caplacizumab up to 30 days after the last PE session.
  Other Names: anti-vWF Nanobody; ALX-0081
  Arms: Caplacizumab
Biological: Placebo — * Subjects received a first i.v. bolus of placebo via push injection within 6 hours to 15 minutes prior to the first PE on study. The first PE on study could either be the very first PE session for the current episode of aTTP (if the subject was randomized prior to the initiation of PE) or the second PE session (if the subject was randomized after a single PE session).
  * The first PE on study was followed by s.c. administration of placebo within 30 minutes after the end of the PE procedure.
  * All subsequent study drug administrations were daily s.c. injections within 30 minutes after the end of the PE procedure (if applicable) or within 24 hours of the previous dose.
  * Subjects received placebo up to 30 days after the last PE session.
  Arms: Placebo

SUMMARY:
This study was a Phase II, single-blind, randomized, placebo-controlled trial to determine whether anti-vWF Nanobody is safe and effective as adjunctive treatment in patients with aTTP.

Patients received either placebo or anti-vWF Nanobody as adjunctive therapy to plasma exchange (PE).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older (adults) or aged 12 to < 18 years (adolescents)
* Male or female subject, willing to accept an acceptable contraceptive regimen
* Subject with a clinical diagnosis of TTP
* Requiring PE (one single PE session prior to randomization into the study was allowed)
* Subject accessible to follow-up
* Subject able to provide signed and dated informed consent and assent (if applicable, for adolescents)

Exclusion Criteria:

* Platelet count ≥ 100,000/µL
* Severe active infection indicated by sepsis (requirement for pressors with or without positive blood cultures)
* Clinical evidence of enteric infection with Escherichia coli 0157 or related organism
* Anti-phospholipid syndrome
* Diagnosis of disseminated intravascular coagulation (DIC)
* Pregnancy or breast-feeding
* Hematopoietic stem cell or bone marrow transplantation-associated thrombotic microangiopathy
* Known with congenital TTP
* Active bleeding or high risk of bleeding
* Uncontrolled arterial hypertension
* Known chronic treatment with anticoagulant treatment that cannot be stopped safely, including but not limited to:

  * vitamin K antagonists
  * heparin or low molecular weight heparin (LMWH)
  * non-acetyl salicylic acid non-steroidal anti-inflammatory molecules
* Severe or life threatening clinical condition other than TTP that would impair participation in the study
* Subjects with malignancies resulting in a life expectation of less than 3 months
* Subjects with known or suspected bone marrow carcinosis
* Subjects who cannot comply with study protocol requirements and procedures
* Known hypersensitivity to the active substance or to excipients of the study drug
* Severe liver impairment, corresponding to grade 3 toxicity defined by the CTCAE scale. For the key liver parameters, this is defined as follows:

  * bilirubin > 3 x upper limit of normal (ULN) (needed to differentiate isolated increase in indirect bilirubin due to hemolysis, this was not an exclusion parameter but disease-related)
  * alanine transaminase (ALT)/ aspartate transaminase (AST) > 5 x ULN
  * alkaline phosphatase (ALP) > 5 x ULN
  * gamma-glutamyl transpeptidase (GGT) > 5 x ULN
* Severe chronic renal impairment, as defined by glomerular filtration rate < 30 mL/min

Note that the use of another investigational drug or device within 30 days prior to screening was not allowed. Participation in non-interventional/observational studies and registries during the study period was allowed. Participation in another clinical study was not allowed until the end of the follow-up period or within 30 days after the last study treatment in case of early subject withdrawal from the study. Subjects who had already participated in the current study and had either completed the study per protocol or had discontinued prematurely, were not allowed to be re-included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Ablynx NV
Locations (51):
- United States (13):
  - Investigator Site, Los Angeles, California
  - Investigator Site, Washington D.C., District of Columbia
  - Investigator Site, Atlanta, Georgia
  - Investigator Site, St Louis, Missouri
  - Investigator Site, New York, New York
  - Investigator Site, Rochester, New York
  - Investigator Site, Valhalla, New York
  - Investigator Site, Durham, North Carolina
  - Investigator Site, Winston-Salem, North Carolina
  - Investigator Site, Columbus, Ohio
  - Investigator Site, Pittsburgh, Pennsylvania
  - Investigator Site, Dallas, Texas
  - Investigator Site, Salt Lake City, Utah
- Australia (4):
  - Investigator Site, Garran, Australian Capital Territory
  - Investigator Site, Liverpool
  - Investigator Site, Melbourne
  - Investigator Site, Woolloongabba
- Austria (2):
  - Investigator Site, Graz
  - Investigator Site, Vienna
- Belgium (4):
  - Investigator Site, Antwerp
  - Investigator Site, Brussels
  - Investigator Site, Leuven
  - Investigator Site, Namur
- Investigator Site, Sofia, Bulgaria
- Investigator Site, Caen, France
- Germany (9):
  - Investigator Site, Ulm, Baden-Wurttemberg
  - Investigator Site, Aachen
  - Investigator Site, Berlin
  - Investigator Site, Cologne
  - Investigator Site, Dortmund
  - Investigator Site, Hanover
  - Investigator Site, Mainz
  - Investigator Site, Mannheim
  - Investigator Site, München
- Israel (3):
  - Investigator Site, Haifa
  - Investigator Site, Jerusalem
  - Investigator Site, Petah Tikva
- Italy (5):
  - Investigator Site, Catania
  - Investigator Site, Foggia
  - Investigator Site, Milan
  - Investigator Site, Reggio Emilia
  - Investigator Site, Rome
- Investigator Site, Bucharest, Romania
- Spain (3):
  - Investigator Site, Badalona
  - Investigator Site, Seville
  - Investigator Site, Valencia
- Switzerland (3):
  - Investigator Site, Bern
  - Investigator Site, Lausanne
  - Investigator Site, Zurich
- United Kingdom (2):
  - Investigator Site, Liverpool
  - Investigator Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Peyvandi F, Cataland S, Scully M, Coppo P, Knoebl P, Kremer Hovinga JA, Metjian A, de la Rubia J, Pavenski K, Minkue Mi Edou J, De Winter H, Callewaert F. Caplacizumab prevents refractoriness and mortality in acquired thrombotic thrombocytopenic purpura: integrated analysis. Blood Adv. 2021 Apr 27;5(8):2137-2141. doi: 10.1182/bloodadvances.2020001834. PMID 33881463
- [Derived] Peyvandi F, Scully M, Kremer Hovinga JA, Cataland S, Knobl P, Wu H, Artoni A, Westwood JP, Mansouri Taleghani M, Jilma B, Callewaert F, Ulrichts H, Duby C, Tersago D; TITAN Investigators. Caplacizumab for Acquired Thrombotic Thrombocytopenic Purpura. N Engl J Med. 2016 Feb 11;374(6):511-22. doi: 10.1056/NEJMoa1505533. PMID 26863353
- [Derived] Holz JB. The TITAN trial--assessing the efficacy and safety of an anti-von Willebrand factor Nanobody in patients with acquired thrombotic thrombocytopenic purpura. Transfus Apher Sci. 2012 Jun;46(3):343-6. doi: 10.1016/j.transci.2012.03.027. Epub 2012 Apr 3. PMID 22475545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with aTTP were recruited from 11 countries in Europe, Australia, Asia and United States (US). Only adults were recruited; no adolescent patients were enrolled, although the trial was open for adolescent patients. A total of 75 patients were included in the trial.
Pre-assignment Details: 76 subjects were screened, 75 subjects were randomized (= Intent-to-treat [ITT] population): 36 in the ALX-0081 group, 39 in the placebo group.
Groups:
- Caplacizumab: Caplacizumab:
  * Subjects received a first i.v. bolus of 10 mg (filled at 5 mg/mL) caplacizumab via push injection within 6 hours to 15 minutes prior to the first PE on study. The first PE on study could either be the very first PE session for the current episode of aTTP (if the subject was randomized prior to the initiation of PE) or the second PE session (if the subject was randomized after a single PE session).
  * The first PE on study was followed by s.c. administration of 10 mg study drug within 30 minutes after the end of the PE procedure.
  * All subsequent study drug administrations were daily s.c. injections within 30 minutes after the end of the PE procedure (if applicable) or within 24 hours of the previous dose.
  * Subjects received caplacizumab up to 30 days after the last PE session.
Period: Overall Study
Arm/Group | Caplacizumab | Placebo
Started | 36 | 39
Received Study Drug | 35 | 37
Completed | 20 | 21
Not Completed | 16 | 18
Not completed — Study terminated by Sponsor | 9 | 10
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Diagnosed as non-TTP patient | 0 | 1
Not completed — Participated in other clinical trial | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caplacizumab | Placebo | Total
Number analyzed (Participants) | 36 | 39 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 38 | 73
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.7) | 42.5 (13.18) | 41.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 12 | 19 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 32 | 34 | 66
  Race/Ethnicity: Black | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time-to-response of Treatment Defined by a Confirmed Recovery of Platelets ≥ 150,000/µL
Description: Time-to-response, defined by the achievement of platelet count response, confirmed at 48 hours after the initial reporting of this response. Platelet response was defined as recovery of platelets ≥ 150,000/µL.
  This response had to be confirmed at 48 hours after the initial reporting of platelet recovery ≥ 150,000/µL by a de novo measure of platelets ≥ 150,000/µL and lactate dehydrogenase (LDH) ≤ 2x upper limit of normal (ULN) (i.e., 'confirmed platelet response').
Time Frame: From the day of first study drug administration up to 30 days after first study drug administration
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
days
  YES - One PE session prior to randomization | 2.4 [1.9 to 3] | 4.3 [2.9 to 5.7]
  NO - No PE session prior to randomization | 3 [2.7 to 3.9] | 4.9 [3.2 to 6.6]
Statistical Analysis 1: Comparison: Caplacizumab vs Placebo; The primary analysis consisted of a Kaplan-Meier analysis with time-to-response as endpoint and treatment group as the independent variable and stratified for absence/presence of one PE session prior to randomization; Test type: Superiority; p = 0.005, Stratified log-rank test — Caplacizumab was compared to placebo using a one-sided log-rank test in order to assess superiority at 2.5% significance level; Hazard Ratio (HR) = 2.2, 95% CI 2-sided [1.28 to 3.78] — The HR was estimated from a Cox proportional Hazards regression model with presence (yes) / absence (no) of 1 PE session prior to randomization as covariate

2. Secondary Outcome: Number and Percentage of Subjects With Complete Remission Following Initial Daily Plasma Exchange (PE)
Description: Number and percentage of subjects with complete remission (defined as confirmed platelet count response and absence of exacerbation) following initial daily PE.
Time Frame: From the day of first study drug administration up to 30 days after first study drug administration
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
Participants | 29 | 18

3. Secondary Outcome: Number and Percentage of Subjects With Exacerbations of TTP
Description: Number and percentage of subjects with exacerbations of TTP (defined as recurrent thrombocytopenia following a confirmed platelet count response and requiring a re-initiation of daily PE treatment after ≥ 1 day but ≤ 30 days of end of daily PE treatment.
  Time to first exacerbation of TTP was also examined as part of this end point analysis; the median time to first exacerbation could not be determined because of the small number of events.
Time Frame: Within 30 days of last day of initial daily PE
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
Participants | 3 | 11

4. Secondary Outcome: Number and Percentage of Subjects With Relapse of TTP
Description: Number and percentage of subjects with relapse of TTP (defined as de novo TTP event that occurred later than 30 days after the last daily PE) was evaluated.
Time Frame: Later than 30 days after the last daily PE
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
Participants | 11 | 3

5. Secondary Outcome: Number of Daily PE Sessions During the Initial Daily PE Period
Description: Number of daily PE sessions during the initial daily PE period which could include more than 1 PE per day was evaluated.
Time Frame: During the initial daily PE period, with a median (min, max) duration of exposure to study drug of 6 (2, 36) days
Population: Number of subjects from the ITT Population with data available
Measure: Mean (Standard Deviation); unit: PE sessions
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
PE sessions | 6.7 (3.69) | 8.4 (6.74)

6. Secondary Outcome: Total Volume of Plasma Administered During the Initial Daily PE Period
Description: The total volume of plasma administered during the initial daily PE period was measured.
Time Frame: During the initial daily PE period, with a median (min, max) duration of exposure to study drug of 6 (2, 36) days
Population: Number of subjects from the ITT Population with data available
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 34 | 37
mL | 22481.8 (15914.85) | 28358.4 (21344.16)

7. Secondary Outcome: Number of Days With at Least One PE Administration During the Total Course of the Study
Description: Number of days for PE was evaluated. This implies the number of days with at least one PE administration during the total course of the study.
Time Frame: During the total course of the study (from Screening till the 12-month follow-up [FU] visit)
Population: Number of subjects from the ITT Population with data available
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
days | 11.8 (7.43) | 12.6 (9.15)

8. Secondary Outcome: The Maximum Number of Consecutive Days Per Subject Where There Was no Interruption of PE During the Initial Daily PE Period
Description: The maximum number of consecutive days per subject where there was no interruption of PE during the initial daily PE period.
Time Frame: During the initial daily PE period, with a median (min, max) duration of exposure to study drug of 6 (2, 36) days
Population: Number of subjects from the ITT Population with data available
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
days | 6.6 (3.35) | 8.1 (6.46)

9. Secondary Outcome: Resolution of Non-focal Neurological Symptoms
Description: Resolution of non-focal neurological symptoms as defined by neurocognitive function at complete remission, measured by a Computerised Neuropsychological Test Battery(CNTB) (adults only). The CNTB included 6 modules: word list learning and selective reminding (WLL/SR), choice reaction time (CRT), visual memory (VMEM), simple reaction time (SRT), working memory (WMEM), and word list learning and delayed recall (WLL/DR). The 6 tasks are rated as a percentage correct (for CRT and SRT, the percentage correct corresponds to the percentage hits) and the mean score from these provides the CNTB summary score (range: 0-100). A higher CNTB summary score indicates better neuropsychological functioning.
Time Frame: From Baseline till the 12-month FU visit
Population: The Computerized Neuropsychological Test Battery (CNTB) was completed by a low proportion of subjects with baseline data available for only 3 subjects in the caplacizumab and 4 subjects in the placebo group and 12 month post-discharge data available for 10 and 6 subjects, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
score on a scale
  Baseline: number analyzed (Participants) | 3 | 4
  Baseline | 66.76 (11.88) | 49.62 (12.91)
  12 months post discharge: number analyzed (Participants) | 10 | 6
  12 months post discharge | 62.10 (12.06) | 58.36 (10.23)

10. Secondary Outcome: Number of Participants With Resolution of TTP-related Signs or Symptoms
Description: Resolution or improvement (improvement of ≥ 1 grade in the Common Terminology Criteria for Adverse Events [CTCAE] v4.0 scale) of TTP-related signs and symptoms as captured on physical examination and as adverse events. This endpoint was only evaluated for "resolution".
Time Frame: End of daily PE treatment period (median [min, max] duration of exposure to study drug of 6 [2, 36] days), end of study treatment period (median [min, max] duration of exposure to study drug of 36.5 [2, 90] days) and at 1 month follow-up
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
Participants
  End of daily PE treatment period | 29 | 29
  End of study treatment period | 30 | 33
  At 1 month follow-up | 31 | 27

11. Secondary Outcome: Mortality
Description: Total mortality up to 1 month follow-up.
Time Frame: From the start of the study up to 1 month follow-up
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
Participants | 0 | 2

12. Secondary Outcome: Number of PE Related Adverse Events
Description: Number of PE treatment-related adverse events (AEs).
Time Frame: From the start of the study up to 1 month follow-up
Population: ITT Population
Measure: Number; unit: adverse events
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
adverse events | 72 | 44

13. Secondary Outcome: Number and Percentage of Subjects With PE Related AEs
Description: Number and percentage of subjects with PE related AEs.
Time Frame: From the start of the study up to 1 month follow-up
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 36 | 39
Participants | 20 | 20

14. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) by Severity
Description: Number and severity of TEAEs were evaluated. The severity grades of AEs were defined as: mild, moderate, and severe. Note: the numbers listed do not include the TEAEs with missing severity.
Time Frame: From the start of the study up to 1 month follow-up
Population: Safety Population
Measure: Number; unit: adverse events
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
adverse events
  Mild | 348 | 299
  Moderate | 154 | 173
  Severe | 37 | 23

15. Secondary Outcome: Number and Percentage of Subjects With TEAEs by Severity
Description: Number and percentage of subjects with TEAEs by severity. The severity grades of AEs were defined as: mild, moderate, and severe.
Time Frame: From the start of the study up to 1 month follow-up
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
Participants
  Mild | 31 | 36
  Moderate | 27 | 31
  Severe | 18 | 14

16. Secondary Outcome: Number of TEAEs and Their Relationship to Study Drug
Description: Number of TEAEs and their relationship to study drug were evaluated. Relationship of AEs to study drug was: related, possibly related, and unlikely/not related.
Time Frame: From the start of the study up to 1 month follow-up
Population: Safety Population
Measure: Number; unit: adverse events
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
adverse events
  Related | 12 | 6
  Possibly related | 59 | 9
  Unlikely/not related | 486 | 524

17. Secondary Outcome: Number of Participants Who Developed Treatment-emergent Anti-Drug Antibodies (ADA)
Description: The development of anti-drug antibodies (ADA) was monitored from the start of the study until last follow-up visit.
Time Frame: From the start of the study until last follow-up visit
Population: Number of subjects from the Safety Population with data available
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 32 | 30
Participants | 3 | 0

18. Secondary Outcome: Plasma Concentrations of Caplacizumab
Description: The concentration of caplacizumab in plasma was determined at different time points. pharmacokinetics (PK) Population: the PK Population consisted of all subjects who received the study drug and for whom the primary PK data are considered to be sufficient and interpretable.
Time Frame: From the start of the study up to 1 month follow-up (i.e., at Baseline, Days 1 and 2 of daily PE, last day of daily PE, Day 1 after daily PE, Weeks 1, 2, 3, and 4 after daily PE, Days 3 and 7 of FU and at the 1-month FU visit).
Population: PK Population, no PK data were generated for the subjects in the placebo group
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 0
ng/mL
  Baseline | 100 (0) |
  Day 1 of daily PE, 5 - 10 min postdose | 1765.9 (185.04) |
  Day 1 of daily PE, 3 - 6 hours postdose | 450.4 (36.15) |
  Day 1 of daily PE, 8 - 24 hours postdose | 562 (36.8) |
  Day 2 of daily PE, predose | 288 (24.05) |
  Day 2 of daily PE, 1 - 6 hours postdose | 415.8 (24.75) |
  Day 2 of daily PE, 6 - 12 hours postdose | 570.7 (52.22) |
  Day 2 of daily PE, 18 - 24 hours postdose | 489.3 (32.54) |
  Last day of daily PE, predose | 348.4 (38.32) |
  Day 1 after daily PE | 521.9 (31.52) |
  Week 1 after daily PE | 490.6 (36.11) |
  Week 2 after daily PE | 524.9 (39.37) |
  Week 3 after daily PE | 499.6 (35.1) |
  Week 4 after daily PE | 503.4 (31.21) |
  Day 3 of follow-up period | 346.7 (25.43) |
  Day 7 of follow-up period | 162.3 (20.2) |
  1 month follow-up | 100 (0) |

19. Secondary Outcome: Pharmacodynamics (PD): Ristocetin Cofactor (RICO) Activity Over Time
Description: The change from baseline in RICO activity was measured at different time points.
Time Frame: as for outcome 18
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of RICO activity
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
percentage of RICO activity
  Baseline | 76.2 (4.95) | 82.1 (3.76)
  Day 1 of daily PE, post dose | 16.2 (0.72) | 84.4 (6.09)
  Day 2 of daily PE, post dose | 21.4 (3.64) | 94.4 (3.69)
  Last day of daily PE, post dose | 15.4 (0.39) | 118.2 (1.78)
  Day 1 after daily PE | 19.2 (3.94) | 105.2 (4.31)
  Week 1 after daily PE | 15 (0) | 107.3 (3.05)
  Week 2 after daily PE | 18.9 (2.87) | 109.2 (2.8)
  Week 3 after daily PE | 17.4 (2.34) | 104 (3.46)
  Week 4 after daily PE | 15.1 (0.07) | 105.5 (3.59)
  Day 3 of follow-up period | 42.3 (6.33) | 99.1 (4.56)
  Day 7 of follow-up period | 88.3 (4.99) | 99.7 (4.06)
  1 month follow-up | 94.6 (3.78) | 94.7 (5.35)

20. Secondary Outcome: Pharmacodynamics: Von Willebrand Factor Antigen (vWF:Ag) Over Time
Description: The change from baseline in vWF:Ag concentration was measured at different time points.
Time Frame: From the start of the study drug up to 1 month follow-up (i.e., at Baseline, Days 1 and 2 of daily PE, last day of daily PE, Day 1 after daily PE, Weeks 1, 2, 3, and 4 after daily PE, Days 3 and 7 of FU and at the 1-month FU visit).
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of vWF:Ag
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
Percentage of vWF:Ag
  Baseline | 185.1 (15.09) | 204.4 (14.52)
  Day 1 of daily PE, post dose | 120.6 (7.98) | 166.6 (9.24)
  Day 2 of daily PE, post dose | 94.6 (4.83) | 140.2 (6.16)
  Last day of daily PE, post dose | 93.6 (6.01) | 151.2 (14.25)
  Day 1 after daily PE | 86.2 (6.15) | 166 (10.05)
  Week 1 after daily PE | 93.4 (6.4) | 234.9 (20.91)
  Week 2 after daily PE | 115.9 (12.42) | 242.6 (19.43)
  Week 3 after daily PE | 102.4 (6.45) | 224.2 (18.62)
  Week 4 after daily PE | 100.1 (5) | 204.3 (17.08)
  Day 3 of follow-up period | 137.8 (9.32) | 184.1 (13.89)
  Day 7 of follow-up period | 190.2 (12.9) | 190.3 (14.81)
  1 month follow-up | 176.3 (15.63) | 167.2 (15.46)

21. Secondary Outcome: PD: Coagulation Factor VIII Clotting Activity (FVIII:C) Over Time
Description: The change from baseline in FVIII:C concentration was measured at different ime points.
Time Frame: as for outcome 18
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of FVIII:C activity
Arm/Group | Caplacizumab | Placebo
Number analyzed (Participants) | 35 | 37
Percentage of FVIII:C activity
  Baseline | 144.18 (11.14) | 156.8 (12.54)
  Day 1 of daily PE, post dose | 104 (6.95) | 149 (9.16)
  Day 2 of daily PE, post dose | 90.7 (5.49) | 152.9 (9.41)
  Last day of daily PE, post dose | 102.4 (10.91) | 169.5 (17.79)
  Day 1 after daily PE | 116.3 (13.33) | 234.2 (16.05)
  Week 1 after daily PE | 116.4 (11.73) | 296.8 (26.07)
  Week 2 after daily PE | 125.2 (16.88) | 291.1 (18.25)
  Week 3 after daily PE | 106.3 (9.7) | 273.1 (20.35)
  Week 4 after daily PE | 95.8 (6.09) | 249.1 (18.27)
  Day 3 of follow-up period | 146.3 (12.59) | 227.7 (17.32)
  Day 7 of follow-up period | 208.6 (15.54) | 237.5 (15.65)
  1 month follow-up | 212.2 (17.33) | 200.1 (17.11)

ADVERSE EVENTS:
Time Frame: From time of the first study drug administration up to the last follow-up visit (12 months)
Arm/Group | Caplacizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 2/37
Serious Adverse Events (participants affected / at risk) | 20/35 | 19/37
Other Adverse Events (participants affected / at risk) | 33/35 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caplacizumab (N=35) | Placebo (N=37)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 13 (16) | 13 (17)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Retinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertransaminasemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Autoantibody test (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caplacizumab (N=35) | Placebo (N=37)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 8 (34)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac disorder (Cardiac disorders) | 2 (3) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Diplopia (Eye disorders) | 1 (2) | 2 (2)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 4 (27)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (4)
Constipation (Gastrointestinal disorders) | 7 (8) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 6 (10) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 5 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (20) | 10 (12)
Paraesthesia oral (Gastrointestinal disorders) | 4 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (11) | 7 (9)
Asthenia (General disorders) | 1 (1) | 6 (8)
Catheter site pain (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 6 (10) | 5 (6)
Injection site bruising (General disorders) | 0 (0) | 2 (2)
Injection site hemorrhage (General disorders) | 3 (6) | 1 (1)
Local swelling (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (5) | 0 (0)
Edema peripheral (General disorders) | 2 (3) | 3 (5)
Pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 6 (6)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (6) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (8) | 2 (2)
Transfusion reaction (Injury, poisoning and procedural complications) | 4 (8) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 3 (5) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 3 (3)
Brain natriuretic peptide increased (Investigations) | 2 (2) | 1 (2)
C-reactive protein increased (Investigations) | 2 (3) | 0 (0)
Hemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Haptoglobin decreased (Investigations) | 2 (2) | 1 (1)
Neutrophil count increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 3 (11)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 5 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (6) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 9 (18) | 8 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (6) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 7 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Disturbance in attention (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 3 (3)
Headache (Nervous system disorders) | 11 (19) | 10 (26)
Migraine (Nervous system disorders) | 2 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 7 (13) | 8 (14)
Syncope (Nervous system disorders) | 1 (1) | 2 (4)
Transient ischemic attack (Nervous system disorders) | 2 (3) | 1 (2)
Tremor (Nervous system disorders) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 3 (3) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (5) | 5 (7)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Disorientation (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 5 (8)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (16) | 4 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (6) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (6) | 3 (5)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 4 (4) | 4 (4)
Hypertension (Vascular disorders) | 5 (6) | 6 (7)
Hypotension (Vascular disorders) | 4 (4) | 2 (2)
Phlebitis (Vascular disorders) | 2 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was stopped prematurely before meeting its enrollment target. The study is not considered to have been terminated as sites were requested to perform the assessments until 1-month follow-up if they had subjects in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any results from this study will be according to the principles of the Declaration of Helsinki, in particular point 30, and will require prior review and written agreement of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2013-06-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT01151423/Prot_000.pdf
  • Statistical Analysis Plan (2013-12-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT01151423/SAP_001.pdf